CLINICAL TRIAL: NCT00619944
Title: Lumefantrine Pharmacokinetics When Administered as a Fixed Dose Combination With Artemether in HIV Positive Patients on Lopinavir/Ritonavir
Brief Title: Drug Interaction Study Between Lumefantrine and Lopinavir/Ritonavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Concepta Merry, Infectious Diseases Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CPR 003
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections
Keywords: HIV; lumefantrine; lopinavir; Africa; Antimalarials; treatment naïve
MeSH Terms: conditions — HIV Infections | interventions — Artemether, Lumefantrine Drug Combination; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lumefantrine lopinavir drug interaction arm
  Interventions: Drug: Lumefantrine - lopinavir/ritonavir drug interaction
- 2 (Active Comparator): lumefantrine only arm
  Interventions: Drug: Lumefantrine only arm

INTERVENTIONS:
Drug: Lumefantrine - lopinavir/ritonavir drug interaction — Lumefantrine 480 mg co-formulated with artemether 80 mg administered as single dose to HIV-positive adults receiving lopinavir/ritonavir 400 mg/100 mg twice daily
  Other Names: Coartem tablets; Kaletra/Aluvia tablets
  Arms: 1
Drug: Lumefantrine only arm — Lumefantrine 480 mg co-formulated with artemether 80 mg administered as a single dose to antiretroviral naive HIV-positive patients
  Other Names: Coartem tablets
  Arms: 2

SUMMARY:
With the roll out of antiretroviral therapy (ARV) for HIV across sub-Saharan Africa an unprecedented number of people will be commencing lifelong therapy. Current estimates are that 5-6 million people in sub-Saharan Africa require ART. At the same time, the World Health Organization (WHO) Roll Back Malaria campaign is aggressively promoting the use of artemether/lumefantrine as first-line therapy for malaria in this setting. Many patients in this setting have already become resistant to first-line ARV and have moved onto lopinavir/ritonavir (Kaletra) based second-line regimens. Kaletra is a potent inhibitor of Cytochrome P450 3A4 (CYP 3A4), an enzyme responsible for the metabolism of many drugs which is found predominantly in the liver and the gut. Lumefantrine, and to a lesser extent artemether, is extensively metabolized by CYP 3A4. Therefore when given to a patient already taking Kaletra for HIV, it is likely that elevated levels of these drugs in the patient will result. There is some concern that lumefantrine may be cardiotoxic due to its structural similarity to halofantrine which is known to cause irregular heart rhythms. This has not been borne out as yet in any studies performed with lumefantrine, however it is not known what levels will be achieved in patients when it is administered with a protease inhibitor such as Kaletra. The WHO has not addressed this issue in any of its previous policy documents but has identified ARV-antimalarial drug interaction studies as a research priority. This single dose pharmacokinetic (PK) study aims to compare the levels of lumefantrine/artemether that result when it is given to a patient on Kaletra with patients not on any ARV. Data generated by this study will help address this important knowledge gap which has been identified by WHO and others as meriting urgent investigation.

DETAILED DESCRIPTION:
In 2004 there were an estimated 40 million people living with HIV, 95% of whom live in the developing world. It is estimated that 5-6 million of these require antiretroviral therapy (ARV) now, and this number will continue to rise. At the recent G8 summit in Gleneagles, Scotland, a unanimous commitment to Universal Access to ARV by 2010 was made. This will result in an unprecedented number of individuals, predominantly in the developing world, commencing lifelong therapy with ARV. Currently the recommended second-line therapy for ARV is a combination of two nucleoside reverse-transcriptase inhibitors (NRTI) and a protease inhibitor (PI). The most widely recommended PI at this time in sub-Saharan Africa is Kaletra (Abbott Laboratories) which is a combination of lopinavir, a PI, and ritonavir, a PI that is a potent enzyme inhibitor and acts as a pharmacokinetic enhancer for lopinavir. Although Kaletra is highly effective in the treatment of HIV, it is a drug that has significant potential for drug-drug interactions. These are largely due to ritonavir's, and to a lesser extent lopinavir's, potent inhibition of Cytochrome P450 3A4 (CYP 3A4), which can result in dramatically raised levels of any co-administered drug metabolised by this same route.

Unfortunately these same people are also the constant victims of the malaria pandemic. There are at least 300 million acute cases of malaria each year globally, resulting in more than a million deaths, 90% of which occur in Africa. Increasing resistance to anti-malarials such as chloroquine, amodiaquine, fansidar, sulphadoxine-pyrimethamine (SP) in East and West Africa has led the WHO to recommend artemether-lumefantrine (Coartem - Novartis) as first-line therapy for malaria for adults and children. By 2004, fourteen countries in sub-Saharan Africa had adopted this as official policy, with the WHO applying pressure on the rest to follow as part of its Roll Back Malaria Campaign. The WHO's recommendations however makes no specific reference to the use of artemether-lumefantrine in HIV positive patients, particularly in patients who are being treated with ARV, although in it's document "Malaria and HIV/AIDS Interactions and Implications: Conclusions of a Technical Consultation Convened by WHO, 23-25 June, 2004" it states that "additional research on interactions between antiretroviral and antimalarial drugs is urgently needed." Coartem is already being used in sub-Saharan Africa as treatment for malaria in HIV-positive individuals on ARV, and this trend is likely to continue given the lack of explicit guidelines on their concomitant administration.

Lumefantrine and artemether are both extensively metabolized by CYP 3A4. To date, no data exist with regard to the potential interactions of these drugs with PI. This gives rise for concern, in particular in the case of lumefantrine, that patients administered both drugs concurrently are likely to have elevated lumefantrine levels with potential for associated toxicity. Lumefantrine, unlike its predecessor halofantrine, does not seem to prolong the QT interval (which can lead to adverse cardiac events), however there is no data with regard to the potential for adverse events when administered with PI. Given the unknown potential for interactions when co-administered with PI, in association with the massive roll out that is occurring of both these drugs across sub-Saharan Africa and their concomitant use in patients, it is essential that these issues be addressed to inform policy as a matter of urgency.

Preliminary or supportive data:

Artemether is metabolized via CYP 3A4 to dihydroartemisinin (although both compounds have antimalarial activity, dihydroartemisinin has greater potency). Inhibition of CYP 3A4 would reduce dihydroartemisinin but increase artemether and potentially increase the short half-life of artemether (1 - 2 hours). The effects of PI and NNRTI are unclear.

Lumefantrine and halofantrine are extensively metabolized by CYP 3A4. Inhibition of halofantrine metabolism could potentially prolong QT interval; given the narrow therapeutic index of this drug, combination with PI is contraindicated and NVP and EFV should be used with caution. Lumefantrine does not seem to prolong the QT interval and is much safer than halofantrine. In a single-dose study in combination with ketoconazole, a potent inhibitor of CYP 3A4, lumefantrine Cmax and AUC were doubled but no clinically significant QT effects were noted. Nevertheless, the Novartis Drug Monograph for Coartem lists CYP 3A4 inhibitors, including Ketoconazole and PI, under precautions/contraindications, despite stating in the same document that "dose adjustment of coartemether appears to be unnecessary when administered in association with ketoconazole or another potent inhibitor of CYP 3A4 activity." No studies however exist in the literature or are listed in the product monograph addressing the important potential interaction with PI. The WHO and a recent editorial in AIDS identify an urgent need for interaction data and state that studies should be prioritized to address this gap in knowledge. Currently in practice, coartem is being administered to patients in sub-Saharan Africa and WHO policy and guidelines do not address this issue.

Significance of the study:

As outlined in the background, this study is of urgent public health importance in the developing world where ARV and anti-malarials are used concomitantly. There are increasing numbers of HIV patients in Uganda moving on to second-line therapy with Kaletra and these are already being treated with coartem where they can afford it. The consequences of prescribing these drugs concomitantly have not been elucidated. The WHO has made no recommendations to guide treatment in this situation and there are no study data available to guide policy. Data generated by this study would help address this important gap which has been identified by WHO and others as meriting urgent investigation.

Hypothesis:

That administration of the lumefantrine and artemether-containing antimalarial combination therapy (Coartem) to HIV-positive patients receiving lopinavir/ritonavir (Kaletra) results in increased exposure to lumefantrine and/or artemether thus putting the patient at increased risk of toxicity from these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age over eighteen
* Ability to provide full informed written consent
* Confirmed diagnosis of HIV infection

Exclusion Criteria:

* Haemoglobin < 8 g/dl
* HIV RNA (Viral Load) > 400 c/ml (if on antiretroviral therapy)
* Malaria Parasitaemia
* Liver and renal function tests > 3 times the upper limit of normal
* Pregnancy
* Use of known inhibitors or inducers of cytochrome P450 or P-glycoprotein
* Use of herbal medications
* QTc (Rate adjusted QT interval) > 450 ms (men) or > 470 ms (women)
* Intercurrent illness including malaria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
12 hour pharmacokinetics profile of lumefantrine in HIV-positive patients receiving lopinavir/ritonavir | 11 months

SECONDARY OUTCOMES:
Safety and tolerability of lumefantrine/artemether in HIV-positive Ugandan patients receiving lopinavir/ritonavir | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Concepta A. Merry, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Infectious Diseases Institute, Faculty of Medicine, Makerere University, Kampala, Uganda

REFERENCES:
- [Derived] Hoglund RM, Byakika-Kibwika P, Lamorde M, Merry C, Ashton M, Hanpithakpong W, Day NP, White NJ, Abelo A, Tarning J. Artemether-lumefantrine co-administration with antiretrovirals: population pharmacokinetics and dosing implications. Br J Clin Pharmacol. 2015 Apr;79(4):636-49. doi: 10.1111/bcp.12529. PMID 25297720
- [Derived] Byakika-Kibwika P, Lamorde M, Okaba-Kayom V, Mayanja-Kizza H, Katabira E, Hanpithakpong W, Pakker N, Dorlo TP, Tarning J, Lindegardh N, de Vries PJ, Back D, Khoo S, Merry C. Lopinavir/ritonavir significantly influences pharmacokinetic exposure of artemether/lumefantrine in HIV-infected Ugandan adults. J Antimicrob Chemother. 2012 May;67(5):1217-23. doi: 10.1093/jac/dkr596. Epub 2012 Feb 8. PMID 22316571